CLINICAL TRIAL: NCT01222858
Title: Innovative Technology to Improve Patient Adherence to Weight Loss Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5RC1HL100002-02 (NIH)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: Obesity; Primary Care; Internet; Technology; Behavior Modification
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internet Education Program (Active Comparator): Participants receive 12 weekly Internet-based weight loss lessons containing information for modification of diet and activity behaviors.
  Interventions: Behavioral: Diet and Activity Education
- Innovative Technology Intervention (Experimental): Participants receive a 12-week Internet-based eating and activity intervention including multimedia lessons and enhanced self-monitoring of weight loss behaviors with automated feedback.
  Interventions: Behavioral: Diet and Activity Education; Behavioral: Self-monitoring with Feedback

INTERVENTIONS:
Behavioral: Diet and Activity Education — Education about behavioral modification of eating and activity habits for weight loss.
Behavioral: Self-monitoring with Feedback — Participants self-monitor diet and activity behaviors, which are submitted via a website. Automated feedback on the self-monitoring record is provided to participants.
  Arms: Innovative Technology Intervention

SUMMARY:
The proposed project addresses the significant problem of obesity and uses innovative technology to improve adherence to a behavioral weight loss strategies. If the program is effective, it would provide an outstanding resource for physicians to use with their patients and thus would have tremendous clinical impact.

DETAILED DESCRIPTION:
Overweight/obesity is a major health problem that affects over two-thirds of Americans, increases morbidity and mortality and has annual medical costs exceeding $75 billion. Although many Americans indicate that they are trying to lose weight, adherence to weight loss regimens is often poor. Programs are needed that can improve adherence and weight loss for overweight/obese individuals. Physicians play an important role in motivating patients to improve health behaviors and recent reviews suggest that having physicians advise patients to lose weight and then referring patients to an effective program produces the best behavior change and maintenance. The problem, however, is that physicians currently have limited options for such referrals. The challenge for the field is to develop a program to which physicians can refer their overweight/obese patients. The program must be low cost, easily accessible, and must promote adherence to the weight loss regimen and consequently improve weight loss outcomes.

The goal of this Challenge Grant application is to develop and test an innovative web-based program that would provide an accessible and effective approach to enhancing adherence to clinical recommendations for weight loss. If effective, the program would provide an outstanding resource for physicians and their patients and could consequently have important clinical and public health impact.

We propose to develop a program based on our prior research that uses innovative Internet technology to provide a low cost, easily disseminated program that captures two critical elements of effective behavioral weight loss programs-namely, training in key behavioral weight control strategies and increased participant accountability. Patients, referred by their physician for weight loss, will be offered a 12 week program that they can view at their convenience on their computer. The program will use Web-based interactive multi-media approaches for presentation of the behavioral skills and provide a Web-based form for submission of self-monitoring and weight data; to maximize patient accountability, the program will include a system of automated feedback for participants, which comments on their weight loss to date and their performance within several behavioral weight-loss domains, with suggestions tailored to the characteristics and performance of the individual. Periodic reports on the patients' progress will also be sent to the referring physician. We will test this program in a randomized trial with 250 patients referred by their physicians who will be randomly assigned to either Internet Education (Control) (N=125) or to the Innovative Technology program (N=125). Participants in both groups will receive a 12 week Internet program of either basic weight loss education or the Innovative Technology program and will be weighed at the start and end of the 3 month program and at 3 month follow-up. The primary hypothesis is that patients who are assigned to the Innovative Technology program will achieve larger average weight losses than those in the control group over the 12-week program. Secondary hypotheses are that the Innovative technology group will adhere better over the 12-weeks (assessed by log-ins to the web site and self-reported changes in diet and activity) and achieve better weight losses at 6 months than the control group.

The proposed project addresses the significant problem of obesity and uses innovative technology to improve adherence to a behavioral weight loss strategies. If the program is effective, it would provide an outstanding resource for physicians to use with their patients and thus would have tremendous clinical impact.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 25 and 45 kg/m2
2. Referred by their physician because of an obesity-related co-morbidity, such as diabetes, hypertension or metabolic syndrome
3. All ethnic groups will be recruited
4. No health problems that make weight loss or unsupervised exercise unsafe
5. English speaking
6. Have access to a computer and the Internet

Exclusion Criteria:

1. report a heart condition, chest pain during periods of activity or rest, or loss of consciousness
2. are currently pregnant or intend to become pregnant in the next 12 months
3. are planning to move outside of the state within the next 12 months
4. have participated in a study conducted by the Weight Control & Diabetes Research Center in the past 2 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Weight Loss | Baseline, 3-mos, 6-mos
  Amount of weight lost (kg) from initial body weight at study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Rena R. Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States